CLINICAL TRIAL: NCT07205705
Title: Impact of Partially Replacing Wheat With Millets or Bengal Gram Flour in Rotis on Glycemia and Prediabetes Reversal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F.no.2.1/FCDOC/EC/HAO/2022-23; IIRPSG-2025-01-00736 (Other Grant/Funding Number: Indian Council of Mdiecal Research)
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — foxtail millet trypsin inhibitor III

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Wheat
- Intervention Group (Experimental): Wheat + Barnyard millet/ Wheat +Barley/ wheat+ Bengal gram flour
  Interventions: Dietary Supplement: Millet

INTERVENTIONS:
Dietary Supplement: Millet — Wheat + Barnyard millet/ Wheat +Barley/ wheat+ Bengal gram flour
  Arms: Intervention Group

SUMMARY:
There is limited research on the impact of millets on glycemia, and it remains unclear whether partially replacing wheat in rotis with low glycemic index millets or Bengal gram flour offers greater glycemic benefits compared to whole wheat. This approach has the potential to reduce postprandial and overall glycemia, supporting the reversal of prediabetes through dietary modification alone. This study introduces a novel formulation of rotis using 50:50 blends of wheat with either barnyard millet, barley, or Bengal gram flour, aiming to improve glycemic control without compromising taste. Glycemic response is assessed through a combination of meal tolerance tests, continuous glucose monitoring, and a three-month dietary intervention, providing both immediate and long-term data. Additionally, the study includes a comprehensive metabolic evaluation by measuring serum insulin, inflammatory markers, and free fatty acids key indicators in the progression of prediabetes. Conducted as a randomized controlled trial with 80 participants across four arms (20 per arm), the study comprises three phases: Phase I evaluates immediate glycemic response through a meal tolerance test; Phase II uses continuous glucose monitoring over three days to monitor fluctuations in glucose levels; and Phase III, with 140 participants, assesses the long-term impact of the dietary intervention over three months. The primary objectives are to determine the effect of the interventions on glycemic response and HbA1c, with an expected outcome of a 10% reduction in the area under the curve for overall and postprandial glucose in Phases I and II, and a 10% reduction in HbA1c in Phase III.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years
2. Prediabetes as diagnosed on oral glucose tolerance test (OGTT): Fasting blood glucose ≥100mg/dl and <126 mg/dl and/or 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 gram anhydrous oral glucose).

Exclusion Criteria:

1. Acute infections and advanced end-organ damage
2. History of hepatitis or pancreatitis, abnormal liver and renal functions
3. Recent (<3 months) changes in weight (≥5%) and/or weight-changing medications
4. Any known allergy to wheat or any other grain
5. Subjects with uncontrolled hypothyroidism or hypertension
6. On any drug causing weight gain or weight loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
HbA1c (%) | 3 months

SECONDARY OUTCOMES:
fasting glucose mg/dL) and satiety | 3 months

IPD SHARING:
Plan to Share IPD: No